CLINICAL TRIAL: NCT01053403
Title: The Effects of MDMA on Sleep Architecture, Water Homeostasis and Cognitive Function
Brief Title: Study of the Effects of MDMA/Ecstasy on Water Regulation, Sleep, and Cognition.
Acronym: 2C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Pacific Medical Center Research Institute (Other)
Responsible Party: Principal Investigator, John Mendelson, MD, Senior Scientist, California Pacific Medical Center Research Institute
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB# 2009.099-1 (JMen); 5-R01-DA016776 (NIH); 5R01DA016776 (NIH)
Record Dates: First submitted 2010-01-08; First posted 2010-01-21 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: MDMA Discontinuation Syndrome
Keywords: MDMA; Ecstasy; MDMA effect on sleep; MDMA effect on water homeostasis; MDMA effect on neurocognitive function; Recreational Drug Use; Drug Abuse
MeSH Terms: conditions — Recreational Drug Use; Substance-Related Disorders | interventions — N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- MDMA (Active Comparator)
  Interventions: Drug: 3,4-methylenedioxymethamphetamine or Placebo

INTERVENTIONS:
Drug: 3,4-methylenedioxymethamphetamine or Placebo — 1.5mg/kg MDMA or matched Placebo administered during 2 inpatients stays. There are 2 dosing sessions and all subjects will receive MDMA at least one time.
  Other Names: Ecstasy

SUMMARY:
The purpose of this study is to measure the effects of MDMA on sleep, mood, thinking, and how your body retains water. The researchers are interested in the effects that occur a few hours after taking MDMA as well as effects occurring over the next two days. We will study these effects in a standardized, controlled setting at the Clinical and Translational Science Institute (CTSI) Clinical Research Center (CRC) located at San Francisco General Hospital.

The primary hypotheses are:

1. MDMA will induce sleep disruption, as indicated by comprehensive polysomnography, wrist actigraphy, and self-report sleep measures
2. MDMA will alter sodium and water homeostasis by either increasing or blunting the suppression of arginine vasopressin levels and decreasing free water excretion. Effects will be exacerbated by water loading.

Secondary hypotheses:

1. Acutely, MDMA will increase both positive and negative arousal, and to increase sociability but not autonomy.
2. Acutely, MDMA will increase risk-taking and willingness to donate money to others in an economic decision making task.
3. MDMA will decrease the stressful effects of talking about a negatively-valenced autobiographical but will increase recall for details for these episodes.
4. MDMA will increase oxidative stress markers and possible ameliorating factors (e.g., ADMA).
5. The short form of the serotonin transported promoter region will be associated with greater acute and discontinuation effects of MDMA.

DETAILED DESCRIPTION:
This is a placebo-controlled, double-blind, gender balanced, within-subject study on the acute and 24 to 48 hour post dose effects (discontinuation syndrome) of MDMA on sleep architecture, water homeostasis and neurocognitive function. We will define the signs and symptoms of sleep disruption and time course of alterations in ADH levels and neurocognitive function occurring after administration of a single dose of MDMA in experienced users. The immediate effects of MDMA include euphoria and intoxication; at 24 hours after MDMA these positive effects are replaced by lowered mood and lethargy - we refer to these effects as a discontinuation syndrome. The pleasurable effects of MDMA are thought to be due to elevations of serotonin, norepinephrine and dopamine; the mechanisms of post-MDMA depression are unknown but may be due to relative serotonin depletion. Among its many functions serotonin maintains normal sleep architecture. The effects of MDMA discontinuation on sleep architecture will be assessed using comprehensive polysomnography and wrist actigraphy with measures obtained ~36 hours after a single dose of MDMA. Cognitive measurements will explore the acute effects of MDMA. MDMA can produce hyponatremia. In this study we will evaluate the effects of MDMA on ADH release, urine sodium excretion, and the relationship of gender to these effects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women aged 18 to 50 years.
* If female: abstains from heterosexual sex, not of childbearing potential, or reports using an approved contraceptive.
* Experienced with MDMA
* Fluent in English.
* Willing and able to give written consent.
* Healthy without medical contraindications to MDMA administration determined by the following: medical history, physical examination, 12-lead EKG, hematology, blood chemistry, and urinalysis.
* Blood liver transaminase elevations up to 3 times the upper limit of normal.
* If female: negative pregnancy test at screening and at the beginning of each hospital admission.
* Negative urine drug test at screening and prior to each potential MDMA administration.

Exclusion Criteria:

* Current enrollment in a MDMA, alcohol, or other drug treatment program or current legal problems relating to MDMA, alcohol, or other drug use, including awaiting trial or supervision by a parole or probation officer.
* Participants with a past-history of using only low doses of MDMA
* Currently trying to quit MDMA use.
* Current dependence on any other psychoactive drug (including nicotine).
* Significant physical or psychiatric illness that might impair the ability to safely complete the study or that might be complicated by the study drugs, including prior seizures (after age 8) or other active neurological disease or clinically significant abnormalities on physical examination or screening laboratory values.
* Likelihood of needing medications to treat an illness during the study period.
* Body Mass Index > 30 or < 18.
* HIV seropositive by self-report.
* If female: pregnancy or lactation.
* History of serious adverse event or hypersensitivity to MDMA.
* Currently taking any medication other than over-the-counter non-steroidal anti-inflammatories, topical medications, inhaled asthma therapy, and over-the-counter non-sedating antihistamines.
* Male neck size ≥ 17 inches, female neck size ≥ 16 inches
* Modified Mallampati class ≥ 3.
* Recent travel within 3 days to or from a different time zone, other than Mountain Standard Time.
* Any other medical or psychosocial condition that would preclude useful, safe, or consistent participation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Time course, severity, and characteristics of MDMA discontinuation in experienced MDMA users given a known dose of MDMA | 1 hour post dose through 48 hours post dose
Relate observed discontinuation effects to sleep data: polysomnography, wrist actigraphy, and self-report sleep measures. | 1 hour post dose through 48 hours post dose
Assess the acute effects of MDMA on water and sodium homeostasis | 1 hour post dose through 48 hours post dose

SECONDARY OUTCOMES:
Document the acute effects of MDMA on self-reported measures, including positive and negative arousal, autonomy, and sociability. | 1 hour post dose through 48 hours post dose
Document the acute effects of MDMA on behavioral measures of economic decision making. | 1 hour post dose through 48 hours post dose
Document the acute effects of MDMA on autobiographical speech and memory | 1 hour post dose through 48 hours post dose
Measure the effects of MDMA on ADMA | 1 hour post dose through 48 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: John Mendelson, MD, Principal Investigator — CPMC Research Institute
Locations (1):
- CPMC Addiction & Pharmacology Research Laboratory (APRL), San Francisco, California, United States

REFERENCES:
- See also: Clinical Trials at the Addiction & Pharmacology Research Laboratory — http://www.cpmc.org/professionals/research/trials/aprllisting.html